CLINICAL TRIAL: NCT06245239
Title: Using Perfusion Index in Assessment of Postoperative Pain in Children Undergoing Hypospadias Repair Surgery: an Observational Follow up Study.
Brief Title: Perfusion Index in Assessment of Postoperative Pain in Children.
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Yahia Mohammd El-hagagy, lecturer of anesthesia and intensive care, faculty of medicine, Assiut University, Assiut University
Other Study IDs: AIP0294591
Record Dates: First submitted 2024-01-23; First posted 2024-02-07 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group I: children aged < 3years undergoing hypospadias repair surgery.
  Interventions: Device: perfusion index

INTERVENTIONS:
Device: perfusion index — measurement of perfusion index
  Other Names: PI

SUMMARY:
The aim of this study will be to examine the validity of perfusion index in predicting pain and evaluation of its severity in the postoperative period.

DETAILED DESCRIPTION:
* Hypospadias repair is a common surgery that is accompanied with significant postoperative pain. The largest group of children usually undergo this type of surgery are infants and pre-verbal children who cannot verbally report pain, and their treatment depends typically on behavioral and observational tools. Although these tools are valid and reliable measures in assessment of pediatric pain, they are still hindered by their subjectivity, which consequently could result in inadequate pain treatment that in early childhood may lead to negative behavioral and neurophysiological sequalae.

That is why recent studies have focused on developing more objective measures to evaluate pain especially when self-report is not possible.

* Changes in perfusion index(PI) caused by sympathetic stimulation refers to possible correlation between pain and PI which forms the basis of our study proposing that the PI is a non-invasive easy method that can be used in evaluating pain in infants

ELIGIBILITY:
Inclusion Criteria:

1. patients aged <3 years
2. Sex:- both male and female.
3. ASA I-II
4. Informed written consent obtained from parents or guardians of all patients.
5. Undergoing hypospadias repair surgery

Exclusion Criteria:

1. Patients outside the selective age range
2. Parents or guardians refusing to enroll their child in the study.
3. ASA III or VI
4. Children with behavioral changes or physical developmental delay
5. Children treated with sedatives or anticonvulsants.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged<3 years of both sexes undergoing hypospadias repair surgery.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Detection of the validity of Perfusion index in predicting Postoperative pain assessed by FLACC score | The baseline preoperative Perfusion index., The FLACC score along with the corresponding Perfusion index readings, will be recorded postoperatively: upon arrival to the PACU and every 30 minutes for 2 hours, then at 6, 12, 18, 24 hours.
  The FLACC score along with the corresponding Perfusion index readings

CONTACTS AND LOCATIONS:
Overall Officials: Noha yahia Mohammed, MD, Principal Investigator — lecturer of anesthesia, faculty of medicine, Assiut university, Egypt
Locations (1):
- Noha yahia Mohammed, Asyut, Assuit Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No